CLINICAL TRIAL: NCT02441855
Title: Is There a Potential Role for Echocardiography in Adult Patients With Community-Acquired Pneumonia Who Require Hospitalization ? A Pilot Study
Brief Title: Potential Role for Echocardiography in Adult Patients With Community-Acquired Pneumonia
Status: Completed | Type: Observational
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Ozcan Basaran, M.D, Muğla Sıtkı Koçman University
Other Study IDs: Pneumonia
Record Dates: First submitted 2015-05-08; First posted 2015-05-12 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Community-acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- pneumonia: patients with community-acquired pneumonia
  Interventions: Device: echocardiography
- control: patients admitted to emergency department with shortness of breath
  Interventions: Device: echocardiography

INTERVENTIONS:
Device: echocardiography — echocardiography: Left and right ventricular functions and aortic elastic properties.

SUMMARY:
Despite the efficacy of modern treatment, community-acquired pneumonia (CAP) is the the leading cause of death. Prognostic scores have been developed to estimate the risk of adverse outcome. Several serum biomarkers have been also investigated in patients with CAP. A growing number of echocardiographic markers have been evaluated as possible predictors of prognosis in patients with pulmonary and infectious diseases such as sepsis, septic shock, human immunodeficiency virus infection, pulmonary tuberculosis, and chronic obstructive pulmonary disease. As echocardiography is a non-invasive, reliable, cost-effective, and reproducible diagnostic tool to evaluate cardiac function and structures, the investigators aimed to investigate left and right ventricular functions and aortic elastic properties in CAP patients. Furthermore, the investigators also aimed to observe relationships between echocardiographic findings and inflammatory and cardiac serum biomarkers in patients with CAP.

DETAILED DESCRIPTION:
Despite the efficacy of modern treatment, community-acquired pneumonia (CAP) is the the leading cause of death. Prognostic scores, like the CURB-65 (confusion, urea, respiratory rate, arterial blood pressure and age) score and the pneumonia severity index (PSI) have been developed and validated to estimate the risk of adverse outcome and to register a patient with CAP for hospital admission. Serum biomarkers have been also investigated in patients with CAP like Procalcitonin and C-reactive protein. Elevated N-terminal pro-brain natriuretic peptide (NT-proBNP) has been shown to be associated with adverse prognosis in several cardiac conditions and critically ill patients. NT-proBNP is also shown to be important predictor in the emergency department and in hospitalized patients with CAP. A growing number of echocardiographic markers have been evaluated as possible predictors of prognosis in patients with pulmonary and infectious diseases such as sepsis, pulmonary tuberculosis, and chronic obstructive pulmonary disease. Although effects of pneumonia on cardiac structures is theoretically possible due to increased systemic inflammatory activity, prothrombotic conditions, biomechanical stress on coronary arteries, variations in coronary arterial tone, and altered myocardial metabolic balance during infections, the role of transthoracic echocardiography has never been evaluated in patients with CAP. As echocardiography is a non-invasive, reliable, cost-effective, and reproducible diagnostic tool to evaluate cardiac function and structures, the investigators aimed to investigate left and right ventricular functions and aortic elastic properties in CAP patients. Furthermore, the investigators also aimed to observe relationships between echocardiographic findings and inflammatory and cardiac serum biomarkers in patients with CAP.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age

Exclusion Criteria:

* Patients with active pulmonary tuberculosis
* Hospital-acquired pneumonia
* Severely immunocompromised patients
* Patients undergoing chronic dialysis
* Patients sent for ambulatory treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pneumonia group is defined as patients with community acquired pneumonia diagnosis hospitalised through emergency department. The control group will be consisted of consecutive sex- and age-matched patients admitted to the emergency department.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2015-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
the TAPSE value to discriminate patients with pneumonia | 1 month
  the TAPSE (Tricuspid annular plane systolic excursion ) value to discriminate patients with pneumonia

SECONDARY OUTCOMES:
the BNP value to discriminate patients with pneumonia | 1 month
  the BNP (B-type natriuretic peptide) value to discriminate patients with pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Murat Biteker, Assoc. Prof., Study Director — Muğla Sıtkı Koçman University
Locations (1):
- Mugla Sitki Kocman University Education and Research Hospital, Muğla, Turkey (Türkiye)

REFERENCES:
- [Derived] Biteker FS, Biteker M, Basaran O, Dogan V, Ozlek B, Yildirim B, Ozlek E, Celik O. A small pericardial effusion is a marker of complicated hospitalization in patients with community-acquired pneumonia. J Crit Care. 2018 Apr;44:294-299. doi: 10.1016/j.jcrc.2017.11.030. Epub 2017 Nov 23. PMID 29247912
- [Derived] Biteker FS, Basaran O, Dogan V, Caylak SD, Yildirim B, Sozen H. Prognostic value of transthoracic echocardiography and biomarkers of cardiac dysfunction in community-acquired pneumonia. Clin Microbiol Infect. 2016 Dec;22(12):1006.e1-1006.e6. doi: 10.1016/j.cmi.2016.08.016. Epub 2016 Sep 3. PMID 27596535